CLINICAL TRIAL: NCT04493424
Title: An Open-label, Long Term Safety Trial of Spesolimab Treatment in Patients With Palmoplantar Pustulosis (PPP) Who Have Completed Previous BI Spesolimab Trials
Brief Title: A Study to Test Long-term Treatment With Spesolimab in People With Palmoplantar Pustulosis (PPP) Who Took Part in Previous Studies With Spesolimab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0024; 2020-000189-41 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Palmoplantar Pustulosis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Up to 260 weeks
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Spesolimab

SUMMARY:
This study is open to people with palmoplantar pustulosis who took part in previous clinical studies of a medicine called spesolimab. Participants who benefited from spesolimab treatment in the previous studies can join this study.

The purpose of this study is to find out how safe spesolimab is and whether it helps people with palmoplantar pustulosis in the long-term. Participants are in this study for up to 5 years. During this time they visit the study site every month to get spesolimab injections under the skin.

At study visits, doctors check the severity of participants' palmoplantar pustulosis and collect information on any health problems of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent for the current trial 1368-0024, in accordance with ICH-GCP and local legislation prior to admission to the current trial
* Male or female patients who have completed the treatment period in one of the parent trials without premature discontinuation
* Patients who have obtained an individual health benefit, per investigator judgement (e.g. PPP PGA of 0 (clear) or 1 (almost clear) or other clinical improvement), from treatment in the parent trial
* Women of childbearing potential must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly

Exclusion Criteria:

* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Patients who experienced study treatment-limiting adverse events during the parent trial
* Severe, progressive, or uncontrolled condition such as renal, hepatic, haematological, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or signs and symptoms thereof
* Patients with congestive heart disease, as assessed by the investigator
* Patient with a transplanted organ (with exception of a corneal transplant > 12 weeks prior to screening in parent trial) or who have ever received stem cell therapy (e.g., Prochymal)
* Known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease (e.g. splenomegaly)
* Any documented active or suspected malignancy or history of malignancy at screening, except appropriately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix
* Patients who have developed active or severe infective disease and opportunistic infections/infective diseases
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (6):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - University of Missouri Health System, Columbia, Missouri
  - The Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Menter Dermatology Research Institute, Dallas, Texas
  - University of Utah Health, Murray, Utah
- Australia (4):
  - Paratus Clinical Research Woden, Phillip, Australian Capital Territory
  - Westmead Hospital, Westmead, New South Wales
  - Skin Health Institute Inc, Carlton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (2):
  - Brussels - UNIV Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Canada (4):
  - Dr. Irina Turchin PC Inc., Fredericton, New Brunswick
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
- Czechia (3):
  - CCBR Czech a.s., Pardubice
  - Univ. Hospital Kralovske Vinohrady, Prague
  - Sanatorium Prof. Arenebergera, Prague
- France (3):
  - HOP l'Archet, Nice
  - HOP Saint-Louis, Paris
  - HOP Larrey, Toulouse
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
- Hungary (2):
  - University of Pecs, Pécs
  - Markusovszky University Teaching Hospital, Szombathely
- Japan (23):
  - Fujita Health University Hospital, Aichi, Toyoake
  - Tokyo Dental College Ichikawa General Hospital, Chiba, Ichikawa
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Asahikawa Medical University Hospital, Hokkaido, Asahikawa
  - Takagi Dermatological Clinic, Hokkaido, Obihiro
  - Takamatsu Red Cross Hospital, Kagawa, Takamatsu
  - Sagamihara National Hospital, Kanagawa, Sagamihara
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Tohoku University Hospital, Miyagi, Sendai
  - Shinshu University Hospital, Nagano, Matsumoto
  - Okayama University Hospital, Okayama, Okayama
  - University of the Ryukyus Hospital, Okinawa, Nakagami-gun
  - Nakatsu Dermatology Clinic, Osaka, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Osaka University Hospital, Osaka, Suita
  - Shiga University of Medical Science Hospital, Shiga, Otsu
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Teikyo University Hospital, Tokyo, Itabashi-ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Poland (5):
  - Barbara Rewerska Diamond Clinic, Krakow, Krakow
  - Dermoklinika medical center, Lodz, Lodz
  - Independent Public Clin.Hosp.no1 Lublin, Lublin
  - Municipal Hospital Complex in Olsztyn, Olsztyn
  - Dermmedica Sp. z o.o., Wroclaw, Wroclaw
- Russia (3):
  - SBHI Chelyabinsk Reg.Clin.Derma.Dispen., Chelyabinsk
  - LLC "Medical Center Azbuka Zdorovia", Kazan'
  - Dermatovenereological Dispensary #10, St. Petersburg, Saint Petersburg
- South Korea (3):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (2):
  - Royal Devon and Exeter Hospital, Exeter
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a phase II, open-label, single arm, to test the safety and efficacy of long-term treatment with Spesolimab in patients with Palmoplantar Pustulosis (PPP) who took part in previous studies with Spesolimab
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Spesolimab (BI 655130): The patients were administered 600 milligram (mg) Spesolimab (BI 655130) prefilled syringes subcutaneously in thighs or abdomen every 4 weeks for up to 5 years (260 weeks). Patients were to continue the treatment until no longer benefited under the patient opinion or investigator assessment, or withdrawal of consent, whichever occurred first.
Period: Overall Study
Arm/Group | Spesolimab (BI 655130)
Started | 108
Completed | 0
Not Completed | 108
Not completed — Termination of the trial by the sponsor | 89
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set for maintenance treatment (SAF-MT): Included all patients who received at least one dose of the maintenance treatment Spesolimab (BI 655130).
Arm/Group | Spesolimab (BI 655130)
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 39
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 69
  More than one race | 0
  Unknown or Not Reported | 0
Palmoplantar Pustulosis Area and Severity Index (PPP ASI) [Mean (Standard Deviation); unit: Score in a scale] — The PPP ASI is an investigator assessment of the extent and severity of pustular and plaque lesions on the palms and soles. The index is a linear combination of the percent of surface area of skin affected on the palms and soles of the body and the severity of erythema (E), pustules (P) and scaling / desquamation (D), providing a numeric score for the overall PPP disease state, ranging from 0 (best outcome) to 72 (worst outcome).
  Score in a scale | 24.97 (10.93)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as all adverse events (AEs) occurring between start of treatment in this extension trial and the end of its residual effect period. Adverse events that started before first intake of trial medication in the extension trial and deteriorated under treatment during the extension trial were also considered as 'treatment-emergent'.
Time Frame: From first administration of study drug until last administration of study drug + 112 days, up to 869 days.
Population: Treated Set for Maintenance Treatment (TS-MT):
  This patient set included all patients who received at least one dose of the maintenance treatment 600 mg s.c. every 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab (BI 655130)
Number analyzed (Participants) | 108
Participants | 96

2. Secondary Outcome: Percent Change in Palmoplantar Pustulosis Area and Severity Index (PPP ASI) From Baseline in Parent Trial (NCT04015518) at Weeks 48 and 96
Description: Percent change in PPP ASI from baseline in parent trial is reported. The adaptation from Psoriasis Area and Severity Index was used in this trial. The index is a linear combination of the percent of surface area of skin affected on the palms and soles of the body and the severity of erythema (E), pustules (P) and scaling / desquamation (D), providing a numeric score for the overall PPP disease state, ranging from 0 (best outcome) to 72 (worst outcome), calculated as: PPP ASI = [(E+P+D) Area x 0.2 (right palm)] + [(E+P+D) Area x 0.2 (left palm)] + [(E+P+D) Area x 0.3 (right sole)] + [(E+P+D) Area x 0.3 (left sole)]. The weighted sum of the scores obtained for Erythema (E), Pustules (P), desquamation (D) (scaling) were based on a score range from 0: None to 4: Very severe, and the area affected on a score range from 0 (0%) to 6 (90-100%). Percent change was calculated as: (PPP ASI at Week X - PPP ASI at baseline in parent trial)/PPP ASI at baseline in parent trial * 100%.
Time Frame: Week 0 (baseline) and Week 48, Week 96
Population: Safety analysis set for maintenance treatment (SAF-MT) This patient set included all patients who received at least one dose of the maintenance treatment.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Spesolimab (BI 655130)
Number analyzed (Participants) | 108
Percent change
  Week 48: number analyzed (Participants) | 84
  Week 48 | -76.85 (22.63)
  Week 96: number analyzed (Participants) | 31
  Week 96 | -77.58 (18.59)

3. Secondary Outcome: Proportion of Patients With PPP ASI50 Compared to Baseline in Parent Trial (NCT04015518) at Weeks 48, 96
Description: Proportion of patients achieving a 50% decrease in PPP ASI compared to baseline in the parent trial at Weeks 48 and 96 is reported. The calculated index is a linear combination of the percent of surface area of skin affected on the palms and soles of the body and the severity of erythema, pustules and scaling / desquamation, providing a numeric score for the overall PPP disease state, ranging from 0 (best outcome) to 72 (worst outcome), calculated as: PPP ASI = [(E+P+D) Area x 0.2 (right palm)] + [(E+P+D) Area x 0.2 (left palm)] + [(E+P+D) Area x 0.3 (right sole)] + [(E+P+D) Area x 0.3 (left sole)]. The weighted sum of the scores obtained for Erythema (E), Pustules (P), desquamation (D) (scaling) were based on a score range from 0: None to 4: Very severe, and the area affected from 0 (0%) to 6 (90-100%). Proportion was calculated as: Patients with PPP ASI50 at Week X/number of evaluable patients at Week X. Non-response imputation (NRI) was used for missing data imputation.
Time Frame: Week 0 (baseline) and Week 48, Week 96
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Spesolimab (BI 655130)
Number analyzed (Participants) | 108
Proportion of participants
  Week 48: number analyzed (Participants) | 100
  Week 48 | 0.770 [0.678 to 0.842]
  Week 96: number analyzed (Participants) | 41
  Week 96 | 0.683 [0.530 to 0.804]

4. Secondary Outcome: Proportion of Patients With PPP PGA of 0 (Clear) or 1 (Almost Clear) at Week 48, 96
Description: Proportion of patients with PPP PGA of 0 (clear) or 1 (almost clear) is reported. The Palmoplantar Pustulosis Physician Global Assessment (PPP PGA) was used to assess the patient's skin presentation on the palms and soles. The investigator scored the individual components (erythema, pustules and scaling/crusting) from 0 to 4 as clear, almost clear, mild, moderate or severe. The PPP PGA was analyzed as PPP PGA total score including erythema, pustules and scaling, and as PPP PGA pustules score for pustules only. Number of patients with PPP PGA of 0/1 at Week X/number of evaluable patients at Week X was calculated. NRI approach was used for missing data imputation.
  The PPP PGA total score was derived as the mean of all individual components:
  0 = If mean=0, for all three components:
  1. = If 0 < mean <1.5
  2. = If 1.5 <= mean <2.5
  3. = If 2.5 <= mean <3.5
  4. = If mean >=3.5
Time Frame: Week 48 and Week 96
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Spesolimab (BI 655130)
Number analyzed (Participants) | 108
Proportion of participants
  Week 48: number analyzed (Participants) | 100
  Week 48 | 0.720 [0.625 to 0.799]
  Week 96: number analyzed (Participants) | 41
  Week 96 | 0.707 [0.555 to 0.824]

ADVERSE EVENTS:
Time Frame: From first administration of study drug until last administration of study drug + 112 days, up to 869 days.
Description: Safety analysis set for maintenance treatment (SAF-MT): This patient set includes all patients who received at least one dose of the maintenance treatment.
Arm/Group | Spesolimab (BI 655130)
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 19/108
Other Adverse Events (participants affected / at risk) | 77/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab (BI 655130) (N=108)
Cardiac failure chronic (Cardiac disorders) | 1
Tricuspid valve incompetence (Cardiac disorders) | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Paraspinal abscess (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Toxic shock syndrome (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Obesity (Metabolism and nutrition disorders) | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab (BI 655130) (N=108)
Injection site erythema (General disorders) | 20
Injection site induration (General disorders) | 6
Injection site pain (General disorders) | 9
Injection site pruritus (General disorders) | 6
Injection site swelling (General disorders) | 12
Injection site warmth (General disorders) | 6
Pyrexia (General disorders) | 14
COVID-19 (Infections and infestations) | 30
Nasopharyngitis (Infections and infestations) | 16
Upper respiratory tract infection (Infections and infestations) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 11
Headache (Nervous system disorders) | 8
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7
Eczema (Skin and subcutaneous tissue disorders) | 9
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 8

LIMITATIONS AND CAVEATS:
The trial was prematurely discontinued due to the sponsor's (Boehringer Ingelheim) decision to terminate the clinical program studying spesolimab in patients with PPP. This decision was not based on any safety finding in the clinical trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT04493424/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT04493424/SAP_001.pdf